CLINICAL TRIAL: NCT06467864
Title: Predicting Ventilator-associated Lower Respiratory Tract Infection Outcomes Using Sequenced-based Early Microbiological Response: A Multi-center Prospective Study
Brief Title: Predicting Ventilator-associated Lower Respiratory Tract Infection Outcomes Using Sequenced-based Early Microbiological Response
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Shanghai East Hospital of Tongji University (Other); First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-SR-223
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pneumonia, Ventilator-Associated; Respiratory Tract Infections; Prognosis
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Respiratory Tract Infections | interventions — Bronchoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — We will perform bronchoscopy and collect bronchoalveolar lavage fluid (BALF) samples at the time of patient enrollment and three days after the treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bronchoscope — We will perform bronchoscopy and collect bronchoalveolar lavage fluid (BALF) samples at the time of patient enrollment and three days after the treatment.

SUMMARY:
We are using a tool called QtNGS (quantitative targeted amplicon-based next-generation sequencing ) to measure the abundance of local pathogens in patients with ventilator-associated lower respiratory tract infections. We hypothesize that changes in pathogen abundance before and after treatment are related to patient outcomes. This study aims to evaluate the effectiveness of the tool by analyzing the changes in pathogen abundance and exploring the relationship between these changes and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above.
* Previously relied on mechanical ventilation (endotracheal intubation or tracheotomy) for breathing assistance, and the duration of mechanical ventilation was more than 48h.
* Lower respiratory tract infection based on at least two of the followings: abnormal temperature (body temperature greater than 38.5°C or less than 36.5°C), leucocyte count abnormality (leucocyte count greater than 12*10^9/L or less than 4*10^9/L), and the presence of purulent tracheal secretions.

Exclusion Criteria:

* Bronchoscopy and respiratory specimen collection were not performed at screening (Day 1) and after 3 days of treatment (Day 4).
* Refusal of patients or families to participate in the study
* After initial screening, bronchoscopy was performed to obtain BALF for bacterial culture. The results of the culture showed no evidence of infection by study-associated lower respiratory pathogens.

Note: The evidence of infection was defined as a single positive bacterial culture (pathogen quantification ≥10^4 cfu/ml or "++" and more) on Day1. And the study-associated causative pathogens are Pseudomonas aeruginosa, Acinetobacter baumannii, Klebsiella pneumoniae, and Staphylococcus aureus. Additionally, the included patient must have single infection with one of these pathogens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population description specifies individuals diagnosed with Va-LRTI (Ventilator-associated Lower Respiratory Tract Infection) who were enrolled based on culture-confirmed pathogens, including Pseudomonas aeruginosa, Acinetobacter baumannii, Klebsiella pneumoniae, and Staphylococcus aureus.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
28-day Mortality Rate | 28 day after enrollment
  The 28-day mortality rate will be measured to determine the percentage of patients who die within 28 days of study enrollment. This outcome will help assess the effectiveness of QtNGS in evaluating early microbiological response.

CONTACTS AND LOCATIONS:
Locations (1):
- he First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China